CLINICAL TRIAL: NCT01339949
Title: A Double-masked, Sham Controlled, Study to Evaluate the Safety and Effectiveness of Low Voltage Stereotactic Radiosurgery in Wet AMD Patients With Recurrent Leakage Secondary to CNV
Brief Title: Study to Evaluate the Safety and Effectiveness of IRay in Wet Age-related Macular Degeneration (AMD) Patients With Recurrent Leakage Secondary to Choroidal Neovascularisation (CNV)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to withdraw study to pursue others.
Sponsor: Oraya Therapeutics, Inc. (Industry)
Responsible Party: Denis O'Shaughnessy, PhD / VP, Clinical Affairs, Oraya Therapeutics, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLH005
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Wet Age-related Macular Degeneration; Age-related Macular Degeneration; AMD; Wet AMD; Macular Degeneration
Keywords: AMD; wet AMD; Macular Degeneration; wet Age-related Macular Degeneration; Age-Related Macular Degeneration; IRay; radiation; Oraya; Oraya Therapeutics, Inc; Low-voltage stereotactic radiosurgery; radiosurgery; x-ray; Lucentis; external beam radiation
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24 Gy radiation (Experimental)
  Interventions: Device: IRay
- Sham 24 Gy radiation (Sham Comparator)
  Interventions: Device: IRay

INTERVENTIONS:
Device: IRay — low voltage external beam radiosurgery
  Arms: 24 Gy radiation
Device: IRay — low voltage external beam radiosurgery
  Arms: Sham 24 Gy radiation

SUMMARY:
The objective of this study is to confirm the safety and to establish the effectiveness of low voltage external beam radiosurgery using the IRay System for the treatment of subjects with recurrent leakage secondary to neovascular Age-related Macular Degeneration (AMD) as determined by decreasing the number of Lucentis injections required during the first 12 months of the study.

DETAILED DESCRIPTION:
The objective of this study is to confirm the safety and to establish the effectiveness of low voltage external beam radiosurgery using the IRay System for the treatment of subjects with recurrent leakage secondary to neovascular AMD as determined by decreasing the number of Lucentis injections required during the first 12 months of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have neovascular AMD, have received at least 6 prior injections with Lucentis or Avastin and have exhibited one or more of the following:

   * have persisting fluid despite 3 consecutive monthly injections of anti- VEGF, or
   * received 4 prior injections over a 6 month period, or
   * received 8 prior injections over a 12 month period.
2. Subjects must now have the need for further anti-VEGF treatment due to increased fluid or persistent cysts on OCT, or leakage on FA.
3. Subjects must have a total lesion size of ≤12 disc areas and a CNV lesion with the greatest linear dimension of ≤6 mm, but not greater than 3 mm from the center of the fovea to the furthest point on lesion perimeter.
4. Subjects must have signed (and been given) a copy of the informed consent form, and be willing and able to return for scheduled treatment and follow-up examinations for the 3-year duration of the study.
5. Subjects must be at least 50 years of age.
6. Women must be post-menopausal ≥1 year or surgically sterilized, or a pregnancy screen must be performed prior to the study and a reliable form of contraception approved by the investigator must be maintained during the study.
7. Subjects must have best corrected visual acuity of 75 to 25 letters in the study eye and at least 20 letters in the fellow eye.

Exclusion Criteria:

1. CNV due to causes other than AMD, including ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia (spherical equivalent ≥-8 diopters).
2. A globe axial length of <20 mm or >26 mm.
3. Evidence of uncontrolled diabetes as determined by an HbA1c of >6.5% and/or with retinal findings consistent with diabetic retinopathy.
4. Prior or concurrent therapies for age related macular degeneration including submacular surgery, subfoveal thermal laser photocoagulation (with or without photographic evidence), transpupillary thermotherapy (TTT), or ocular photodynamic therapy in the study eye.
5. History of radiation to the head in the region of the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Number of Lucentis injections during first 52 weeks | 52 weeks

SECONDARY OUTCOMES:
Change in mean VA | 52 weeks
Loss/gain of letters of BCVA | week 52

CONTACTS AND LOCATIONS:
Locations (3):
- Università Vita-Salute Istituto Scientifico San Raffaele, Milan, Italy
- United Kingdom (2):
  - King's College Hospital, London
  - Manchester Royal Eye Hospital, Manchester